CLINICAL TRIAL: NCT05239936
Title: Urdu Version of Arthritis Impact Measurement Scales 2 Short Form:Reliability and Validity Study Among Patients With Osteoarthritis
Brief Title: Urdu Version of Arthritis Impact Measurement Scales 2 Short Form:Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00253
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Quality of Life
Keywords: AIMS2 SF; Urdu; OA; ACR

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study ,Investigators will observe the Reliability and Validity of Arthritis Impact Measurement Scale 2 Short Form translated in Urdu language in Pakistani population to check quality of life in patients suffering from Osteoarthritis.

DETAILED DESCRIPTION:
The main aim of this study is to translate and culturally adapt AIMS2 SF into Urdu language and to investigate the reliability and validity of AIMS2 SF in Osteoarthritis patients among Urdu speaking Pakistani population.

The study will be completed in 5 steps such as translation ,synthesis ,back translation ,expert committee review and pre testing. The study will be a cross sectional survey .The result of the study helps to know the validity and reliability of AIMS2 SF in Urdu Version to check the quality of life .The reliability of the scale will be checked through internal consistency and test retest method .Internal consistency will be analyzed through Cronbach's alpha value to estimate whether each item of a scale is appropriate for assessing the underlying concept of its scale with 165 patients will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female Patient age 18 years or older.
2. Diagnosed with OA of the knee , hip and hand .
3. Patients diagnosed according to ACR criteria. 4 - X-RAY scored according to Kellgren and Lawrence Classification.

Exclusion Criteria:

1 - Radiograph not older than 6 months . 2- Age less than 18 are excluded from this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoarthritis is the leading cause of pain and disability and the most common joint disorder in our general population .According to high prevalence due to increasing age it is also increasing in the upcoming years .It causes narrow joint space and degeneration of cartilage
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Arthritis Impact Measurement Scale 2-Short Form | 1st day
  Arthritis Impact Measurement Scale 2-Short Form was designed to study Arthritis outcomes .It is a self administrated ,multidimensional health status assessment tool. Arthritis Impact Measurement Scale 2-Short Form has been extensively validated and shown to be reliable in cross sectional studies and clinical trails

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index | 1st day
  Western Ontario and McMaster Universities Arthritis Index is used in evaluation of hip and knee Osteoarthritis. This is consisting of 24 items which are further divided into 3 subscales. 1-pain (5 items) 2- Stiffness (2 items) 3- Physical Function (17)items

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No